CLINICAL TRIAL: NCT01288625
Title: Prospective, Open-label, Randomized, Control Study of Head and Neck Cancer Radiation Treatment With or Without Amifostine
Brief Title: Prospective Study of Head and Neck Cancer Radiation Treatment With or Without Amifostine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: There were IP availability issues due to which the study could not be started.
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SUN-2011-DP
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Oral Mucositis; Stomatitis
Keywords: Identify whether Cytofos can reduce the incidence and duration of HNC patients' oral mucositis caused by radiotherapy.
MeSH Terms: conditions — Stomatitis | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cytofos group A (Experimental): Amifostine 500 mg sc, qod, 3 times per week Radiation treatment 30 min after amifostine treatment, 1.8-2.0 Gy/day × 30-35 times
  Interventions: Drug: Amifostine; Radiation: Amifostine
- Cytofos group B (Experimental): Amifostine 500mg rinsing wash, qod, 3 times per week Radiation treatment 5 min after amifostine treatment, 1.8-2.0 Gy/day × 30-35 times
  Interventions: Drug: Amifostine; Radiation: Amifostine
- Control group (Active Comparator): Radiation treatment 1.8-2.0 Gy/day × 30-35 times
  Interventions: Drug: Amifostine; Radiation: Amifostine

INTERVENTIONS:
Drug: Amifostine — 500 mg sc, qod, 3 times per week
Radiation: Amifostine — 500mg rinsing wash, qod, 3 times per week

SUMMARY:
The purpose of this study is to compare the incidence of stomatitis when treating with amifostine before radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, male or female
2. Primary treatment of phase I-IVA head and neck cancer patients, identified by histological and pathological diagnosis
3. Postoperative patients should receive radiation treatment in 12 weeks
4. ECOG <2
5. Expected lifetime ≥6months
6. No severe complications (hypertension, CHD, diabetes and psychiatric history, etc.)
7. Not involved in other clinical trials
8. Sign ICF

Exclusion Criteria:

1. ECOG >2
2. Suffered other cancers in the past 5 years
3. Received amifostine treatment in the past 4 weeks
4. Unable to complete treatment or sign ICF because of medical or physical reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Incidence and duration of oral mucositis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang ge, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University